CLINICAL TRIAL: NCT02187302
Title: A Randomized, Phase 2 Study to Assess the Safety and Efficacy of CRLX101 in Combination With Bevacizumab in Patients With Metastatic Renal Cell Carcinoma (RCC) Versus Standard of Care (SOC) (Investigator's Choice)
Brief Title: CRLX101(NLG207) in Combination With Bevacizumab for Metastatic Renal Cell Carcinoma (mRCC) Versus Standard of Care (SOC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLX101-208
Record Dates: First submitted 2014-06-30; First posted 2014-07-11 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: nanopharmaceutical,
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — IT-101; Bevacizumab; Standard of Care; Sorafenib; Sunitinib; Axitinib; pazopanib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRLX101 + bevacizumab (Experimental): CRLX101 in combination with bevacizumab:
  * CRLX101 15 mg/m^2 IV on days 1 and 15 of a 28-day cycle;
  * bevacizumab 10 mg/kg IV on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: CRLX101; Drug: Bevacizumab
- Standard of Care (Active Comparator): Standard of care treatment include one of the following agents to which the patient can have no prior exposure: sorafenib; everolimus; pazopanib; axitinib; bevacizumab; sunitinib, or other approved drug considered by the Medical Monitor to represent an acceptable standard of care therapy
  Interventions: Drug: Standard of Care (Investigator Choice)

INTERVENTIONS:
Drug: CRLX101
  Other Names: NLG207
  Arms: CRLX101 + bevacizumab
Drug: Bevacizumab
  Other Names: Avastin
  Arms: CRLX101 + bevacizumab
Drug: Standard of Care (Investigator Choice)
  Other Names: sorafenib (Nexavar), sunitinib (Sutent), axitinib (Inlyta), pazopanib (Votrient), bevacizumab (Avastin),; everolimus (Afinitor), Other
  Arms: Standard of Care

SUMMARY:
This study to evaluate treatment in patients with metastatic renal cell carcinoma (RCC) which has progressed through 2 to 3 prior lines of therapy, with the investigational drug CRLX101 in combination with bevacizumab compared to treatment with a standard of care therapy. The study will compare which treatment resulted in longer time before progression of the RCC. Patients will be treated and followed for progression of their disease on average for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed renal cell carcinoma of any pathologic subtype.
* Must have unresectable metastatic disease, and have tumor(s) present that is (are) evaluable by the RECIST, v1.1; may have spinal-associated metastases but must have concluded dexamethasone therapy and be evaluated by the Investigator to have stable CNS disease.
* Must have received 2 or 3 prior lines of conventional molecularly targeted therapy
* Must have full recovery from any toxicities from prior therapy CTCAE Grade 1 or less with the exception of Grade 2 alopecia) prior to randomization.
* ECOG performance status 0 or 1.
* Age 18 years and older.
* Life expectancy of at least 3 months.
* Must have normal organ and marrow function reported within 14 days prior to randomization
* Ability to understand and willingness to sign a written informed consent document.
* Able to comply with study visit schedule and assessments.

Exclusion Criteria:

* Any conventional molecularly targeted therapy within 2 weeks or, chemotherapy or radiotherapy within 2 weeks (local) or 4 weeks (systemic) prior to entering the study.
* Failure to recover to grade 1 or less all prior adverse events.
* Any major surgery within 4 weeks of study randomization.
* Any prior treatment with topoisomerase I therapy.
* Prior treatment with any drugs or therapies that will be administered during the course of this trial including CRLX101, any topoisomerase 1 inhibitor, bevacizumab or the conventional molecularly targeted agent intended for use as standard of care treatment.
* Patients receiving any other current investigational therapeutic agent.
* Other active malignancies
* Patients with brain metastasis treated or untreated, or other CNS disease
* Any clinically significant cardiac disease defined as NYHA class III or IV.
* Uncontrolled hypertension
* Uncontrolled concurrent illness
* History of non-healing wounds or ulcers.
* Pregnancy, or inadequate contraception for men or women of childbearing age, or lactating / breast-feeding
* Patients with known HIV or with solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | at least 6 months
  To assess progression free survival (PFS) in patients with clear cell metastatic renal cell carcinoma (RCC) treated with CRLX101 in combination with bevacizumab (CRLX101+bevacizumab) vs. standard of care (SOC) per investigator's choice, as assessed by blinded independent radiological review (IRR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Overall Safety and tolerability (AEs, SAEs, Clinical Laboratory Parameters, Vital Signs, Concomitant Medications) | at least 30 days post last dose of study drug
  AEs will be coded using MedDRA and graded according to CTCAE (v 4.03). The number and percentage of patients with any treatment-emergent AE (TEAE) will be summarized for each treatment group. The number of patients with TEAEs assessed by the Investigator as at least possibly related to treatment will be tabulated. The number of patients with any CTCAE grade ≥ 3 treatment-emergent AE will be tabulated. Serious AEs (SAEs) will also be tabulated.
  For Clinical Laboratory Parameters - Shift tables that present changes from baseline to worst on-study values relative to CTCAE grading will be produced.
  For Vital Signs - By-patient data listings of vital sign measurements will be presented.
  For Concomitant Medications - The use of concomitant medications will be included in by-patient data listings. A summary table of concomitant medications by WHO drug class will also be provided.
Overall survival | on average 12 months after discontinuation of study treatment
  To compare time to death between treatment groups of CRLX101 in combination with bevacizumab compared to SOC.
Objective response rate | at least 6 months
  Evaluate response rates comparing the investigational treatment of CRLX101 in combination with bevacizumab compared to SOC as assessed by blinded IRR as well as by the Investigator
Duration of Response | at least 6 months
  Evaluate time to response comparing the investigational treatment of CRLX101 in combination with bevacizumab compared to SOC as assessed by blinded IRR as well as by the Investigator
PFS | at least 6 months
  To assess PFS in patients with clear cell metastatic RCC treated with CRLX101+bevacizumab vs. SOC per investigator's choice, as assessed at the site level by the Investigator according to RECIST version 1.1
PFS | at least 6 months
  To assess PFS (as assessed at the site level by the Investigator and separately by blinded IRR) in clear cell RCC patients treated with CRLX101+bevacizumab compared to bevacizumab treatment alone

CONTACTS AND LOCATIONS:
Overall Officials: NewLink Genetics, Study Chair — NewLink Genetics Inc
Locations (43):
- United States (38):
  - University of California San Diego, La Jolla, California
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Kaiser Permanente, Honolulu, Hawaii
  - Decatur Memorial Hospital, Decatur, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Ann Arbor Hematoloty-Oncology, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - North Mississippi Hematology and Oncology Associates, Tupelo, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - MD Anderson Cooper Cancer Institute, Voorhees Township, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology, Amarillo, Amarillo, Texas
  - Texas Oncology P.A., Austin, Texas
  - Texas Oncology, Dallas, Dallas, Texas
  - Texas Oncology, El Paso, El Paso, Texas
  - Texas Oncology, Flower Mound, Flower Mound, Texas
  - Texas Oncology, Fort Worth, Fort Worth, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Cancer Center Network of South Texas, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - CAMC Health Education and Research Institute, Charleston, West Virginia
  - St. Vincent Regional Cancer Center CCOP, Green Bay, Wisconsin
- South Korea (5):
  - National Cancer Center, Goyang-si Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severence Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Voss MH, Hussain A, Vogelzang N, Lee JL, Keam B, Rha SY, Vaishampayan U, Harris WB, Richey S, Randall JM, Shaffer D, Cohn A, Crowell T, Li J, Senderowicz A, Stone E, Figlin R, Motzer RJ, Haas NB, Hutson T. A randomized phase II trial of CRLX101 in combination with bevacizumab versus standard of care in patients with advanced renal cell carcinoma. Ann Oncol. 2017 Nov 1;28(11):2754-2760. doi: 10.1093/annonc/mdx493. PMID 28950297